CLINICAL TRIAL: NCT04305587
Title: A Phase 1, Randomized, Double-Blind, Sponsor-Open, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Escalating Oral Doses of PF-07081532 in Adult Participants With Type 2 Diabetes Mellitus
Brief Title: Multiple Escalating Oral Doses Study of PF-07081532 in Adult Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C3991002
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind (investigator- and participant-blind), sponsor-open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Active Obesity (Experimental): Part B
  Interventions: Other: Placebo; Drug: Clopidogrel
- Placebo Obesity (Placebo Comparator): Part B
  Interventions: Other: Placebo; Drug: Clopidogrel
- Active T2DM (Experimental): Parts A and C
  Interventions: Drug: PF-07081532
- Placebo T2DM (Placebo Comparator): Parts A and C
  Interventions: Drug: PF-07081532

INTERVENTIONS:
Drug: PF-07081532 — Investigational Drug once daily for up to 42 days; multiple ascending dose design.
  Arms: Active T2DM; Placebo T2DM
Other: Placebo — Placebo once daily for up to 42 days.
  Arms: Active Obesity; Placebo Obesity
Drug: Clopidogrel — Part B may include a drug-drug interaction study using open-label clopidogrel. Clopidrogrel may be given as two single doses of 75 mg administered on day -2 and day 41.
  Other Names: Plavix
  Arms: Active Obesity; Placebo Obesity

SUMMARY:
This is a randomized, placebo-controlled, double-blind (investigator- and participant-blinded), sponsor-open, dose-escalating study of PF-07081532 in patients with Type 2 diabetes on metformin (Parts A and C). The study may also enroll non-diabetic participants with obesity (Part B). Study participants will receive an investigational product or placebo every day for up to 28 days (Part A) or up to 42 days (Part B, optional; Part C, optional).

The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple oral doses of PF-07081532 in participants with inadequately controlled T2DM on metformin and optionally in non-diabetic obese participants.

ELIGIBILITY:
Key Inclusion Criteria for participants enrolling with T2DM:

* Type 2 Diabetes treated with a stable dose of metformin at least 500 mg per day for at least 2 months prior to screening visit and use of no other medications for glycemic control.
* HbA1c value between 7.0% and 10.5%, inclusive.

Key Exclusion Criterion for participants enrolling with T2DM:

-Type 1 Diabetes or secondary forms of diabetes.

Key Inclusion Criterion for participants enrolling with obesity:

-Obese (as indicated by screening BMI) non-diabetic adults.

Key Exclusion Criterion for participants enrolling with obesity:

--Type 1 or Type 2 Diabetes or secondary forms of diabetes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Qps-Mra, Llc, South Miami, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Buckeridge C, Tsamandouras N, Carvajal-Gonzalez S, Brown LS, Hernandez-Illas M, Saxena AR. Once-daily oral small-molecule glucagon-like peptide-1 receptor agonist lotiglipron (PF-07081532) for type 2 diabetes and obesity: Two randomized, placebo-controlled, multiple-ascending-dose Phase 1 studies. Diabetes Obes Metab. 2024 Aug;26(8):3155-3166. doi: 10.1111/dom.15643. Epub 2024 May 16. PMID 38751362
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 66 participants were assigned to treatment and received at least 1 dose of study intervention; of these, 61 participants completed the blinded treatment. Of the 5 participants who discontinued study treatment, 3 were due to treatment-related adverse events (AEs), and 2 were due to other reasons. One participant discontinued from study due to withdrawal by participant and other 65 participants completed the study.
Groups:
- Placebo Part A: Adult participants with type 2 diabetes mellitus (T2DM) received oral placebo once daily (QD) over 28 days.
- PF-07081532 10 mg Part A: Adult participants with T2DM received oral PF-07081532 10 milligrams (mg) QD over 28 days.
- PF-07081532 30 mg Part A: Adult participants with T2DM received oral PF-07081532 QD titrated from 10 mg to a target dose of 30 mg over 28 days.
- PF-07081532 60 mg Part A: Adult participants with T2DM received oral PF-07081532 QD titrated from 10 mg to a target dose of 60 mg over 28 days.
- PF-07081532 120 mg Part A: Adult participants with T2DM received oral PF-07081532 QD titrated from 10 mg to a target dose of 120 mg over 28 days.
- Placebo Part B: Adult participants with Obesity (without diabetes) received oral placebo QD over 42 days.
- PF-07081532 180 mg Part B: Adult participants with Obesity (without diabetes) received oral PF-07081532 QD titrated from 10 mg to a target dose of 180 mg over 42 days.
- Placebo Part C: Adult participants with T2DM received oral placebo QD over 42 days.
- PF-07081532 180 mg Part C: Adult participants with T2DM received oral PF-07081532 QD titrated from 10 mg to a target dose of 180 mg over 42 days.
Period: Overall Study
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C
Started | 9 | 7 | 8 | 8 | 8 | 3 | 12 | 2 | 9
Completed | 9 | 7 | 8 | 7 | 8 | 3 | 12 | 2 | 9
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants received at least 1 dose of study intervention (PF-07081532 or placebo) and were included in the baseline analysis population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C | Total
Number analyzed (Participants) | 9 | 7 | 8 | 8 | 8 | 3 | 12 | 2 | 9 | 66
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4
  45-64 years | 7 | 3 | 7 | 5 | 8 | 2 | 10 | 2 | 6 | 50
  >=65 years | 1 | 4 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 4 | 4 | 4 | 2 | 5 | 1 | 4 | 31
  Male | 6 | 3 | 4 | 4 | 4 | 1 | 7 | 1 | 5 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 10
  White | 8 | 5 | 7 | 7 | 7 | 3 | 11 | 2 | 6 | 56
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) Continuous [Mean (Standard Deviation); unit: kilogram/meter^2 (kg/m^2)] | 32.5 (4.70) | 37.4 (4.34) | 32.3 (3.10) | 32.1 (5.81) | 32.9 (6.87) | 37.4 (6.77) | 34.6 (3.50) | 25.7 (0.51) | 31.5 (3.65) | 33.3 (4.99)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Treatment-Related Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An serious adverse event (SAE) was defined as an AE: 1. resulting in death, 2. was life-threatening, 3. required inpatient hospitalization or prolongation of existing hospitalization, 4. resulted in persistent disability, 5. was a congenital anomaly/birth defect, or considered to be an important medical event. Treatment-related AE was any untoward medical occurrence attributed to study intervention in a participant who received study intervention. Treatment-emergent are events between first dose of study intervention and up to 28-35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose up to 28-35 days after last administration of study intervention (that is a maximum of 63 days from first dose for Part A and a maximum of 77 days from first dose for Part B and Part C)
Population: The population for this outcome measure included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C
Number analyzed (Participants) | 9 | 7 | 8 | 8 | 8 | 3 | 12 | 2 | 9
Participants
  Treatment-related AEs | 5 | 2 | 6 | 6 | 8 | 2 | 11 | 2 | 9
  Treatment-related SAEs | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Participants with laboratory abnormalities with ≥2 occurrences (without regard to baseline abnormality) that met pre-specified criteria were High-density lipoprotein (HDL) Cholesterol <0.8✕ lower limit of normal (LLN); Bicarbonate <0.9✕LLN; Calcitonin>1.0✕upper limit of normal (ULN); Triglycerides >1.3✕ULN; Aspartate Aminotransferase >3.0✕ULN; Low-density lipoprotein (LDL) Cholesterol >1.2✕ULN; Urine Glucose ≥1; Urine Ketones ≥1; Urine Leukocyte Esterase ≥1; Urine Leukocytes ≥20; Urine Hyaline Casts >1; Urine Hemoglobin ≥1; and Urine Nitrite ≥1.
Time Frame: From Baseline to 7-14 days following last dose administration (that is a maximum of 42 days from baseline for Part A and a maximum of 56 days from baseline for Part B and Part C)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8 | 3 | 12 | 2 | 9
Participants
  HDL Cholesterol (mg/dL) <0.8✕LLN: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 3 | 12 | 2 | 8
  HDL Cholesterol (mg/dL) <0.8✕LLN | 2 | 0 | 3 | 2 | 1 | 1 | 1 | 1 | 2
  Bicarbonate (milliequivalents per liter [Meq/L]) <0.9✕LLN | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Calcitonin (pg/mL) >1.0✕ULN: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 3 | 12 | 2 | 8
  Calcitonin (pg/mL) >1.0✕ULN | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
  Triglycerides (mg/dL) >1.3✕ULN: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 3 | 12 | 2 | 8
  Triglycerides (mg/dL) >1.3✕ULN | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (U/L) >3.0✕ULN | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
  LDL Cholesterol (mg/dL) >1.2✕ULN: number analyzed (Participants) | 8 | 7 | 8 | 7 | 7 | 3 | 12 | 2 | 8
  LDL Cholesterol (mg/dL) >1.2✕ULN | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
  Urine Glucose ≥1 | 3 | 1 | 2 | 2 | 3 | 0 | 0 | 1 | 1
  Urine Ketones ≥1 | 0 | 0 | 1 | 1 | 3 | 0 | 3 | 0 | 0
  Urine Leukocyte Esterase ≥1 | 1 | 1 | 3 | 1 | 1 | 0 | 2 | 0 | 3
  Urine Leukocytes (/high power field [HPF]) ≥20: number analyzed (Participants) | 4 | 4 | 6 | 4 | 5 | 3 | 8 | 0 | 6
  Urine Leukocytes (/high power field [HPF]) ≥20 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0
  Urine Hyaline Casts (/low power field [LPF]) >1: number analyzed (Participants) | 1 | 2 | 2 | 1 | 3 | 0 | 2 | 0 | 1
  Urine Hyaline Casts (/low power field [LPF]) >1 | 0 | 2 | 2 | 1 | 3 | 0 | 1 | 0 | 1
  Urine Hemoglobin ≥1 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0
  Urine Nitrite ≥1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Number of Participants With Vital Signs Abnormalities
Description: Vital signs (pulse rate, systolic and diastolic blood pressure) were obtained with participant in the supine position. The pre-specified categorical analysis criteria in vital signs, were supine systolic blood pressure < 90 millimeters of mercury (mmHg), supine systolic blood pressure increase/decrease from baseline ≥ 30mmHg; supine diastolic blood pressure <50 mmHg, supine diastolic blood pressure increase/decrease from baseline ≥ 20mmHg; pulse rate <40 beats per minute (bpm) or >120 bpm.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C
Number analyzed (Participants) | 9 | 7 | 8 | 8 | 8 | 3 | 12 | 2 | 9
Participants
  Supine Systolic Blood Pressure (mmHg) - Value <90mmHg | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
  Supine Systolic Blood Pressure (mmHg) - Change ≥ 30mmHg increase | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 0
  Supine Systolic Blood Pressure (mmHg) - Change ≥ 30mmHg decrease | 2 | 1 | 2 | 4 | 3 | 0 | 0 | 0 | 2
  Supine Diastolic Blood Pressure (mmHg) - Value <50 mmHg | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) - Change ≥ 20mmHg increase | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0
  Supine Diastolic Blood Pressure (mmHg) - Change ≥ 20mmHg decrease | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
  Pulse Rate (bpm) - Value <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse Rate (bpm) - Value >120 bpm | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG)
Description: The pre-specified categorical analysis criteria in ECG, were PR interval: value ≥ 300 milliseconds (msec), percentage change ≥ 25/50%; QRS duration: value ≥140 msec, percentage change ≥ 50%; QTcF interval: 450 < value ≤ 480 msec, 480 < value ≤ 500 msec, value >500 msec, and 30<change ≤ 60 msec, change >60 msec.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C
Number analyzed (Participants) | 9 | 7 | 8 | 8 | 8 | 3 | 12 | 2 | 9
Participants
  PR Interval (msec) - Value ≥300 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Interval (msec) - %Change ≥ 25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration (msec) - Value ≥140 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  QRS Duration (msec) - %Change ≥ 50% | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (msec) - 450 < Value ≤ 480 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (msec) - 480 < Value ≤ 500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (msec) - Value >500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTcF Interval (msec) -30 < Change ≤ 60 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
  QTcF Interval (msec) -Change >60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Area Under the Curve From Time 0 to 24 Hours (AUC24) Post Dose for PF-07081532
Description: AUC24 is defined as area under the concentration-time profile from time 0 to 24 hours using Linear/Log trapezoidal method.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24 hours post-dose on Days 1 and 28 for Part A, on Days 1 and 42 for Part B and Part C
Population: The population for this outcome measure included all randomized participants who received at least 1 dose of PF-07081532 and had at least 1 of the pharmacokinetics (PK) parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part B | PF-07081532 180 mg Part C
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 9
nanogram*hour/milliliter (ng*hr/mL)
  AUC24 (Day 1) | 15530 (15) | 14430 (25) | 17220 (34) | 15100 (42) | 14340 (21) | 14560 (35)
  AUC24 (Day 28 or 42) | 26380 (23) | 78930 (20) | 177000 (58) | 265400 (62) | 521300 (38) | 496500 (44)

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for PF-07081532
Description: Cmax is defined as maximum plasma concentration observed directly from data.
Time Frame: as for outcome 5
Population: The population for this outcome measure included all randomized participants who received at least 1 dose of PF-07081532 and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part B | PF-07081532 180 mg Part C
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 9
nanogram/milliliter (ng/mL)
  Cmax (Day 1) | 1599 (17) | 1518 (35) | 1699 (27) | 1548 (37) | 1531 (23) | 1587 (21)
  Cmax (Day 28 or 42) | 2263 (19) | 5631 (26) | 12860 (51) | 18520 (47) | 35000 (37) | 30600 (33)

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-07081532
Description: Tmax is defined as time for Cmax observed directly from data as time of first occurrence.
Time Frame: as for outcome 5
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part B | PF-07081532 180 mg Part C
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 9
hour
  Tmax (Day 1) | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 2.00 [1.00 to 4.00] | 1.00 [0.50 to 6.00] | 1.50 [0.50 to 4.00] | 1.00 [1.00 to 4.00]
  Tmax (Day 28 or 42) | 2.00 [2.00 to 4.00] | 4.00 [1.00 to 12.00] | 4.00 [1.00 to 10.00] | 4.00 [4.00 to 12.00] | 4.00 [1.00 to 12.00] | 8.00 [6.00 to 12.00]

8. Secondary Outcome: Time Measured for the Plasma Concentration to Decrease by One-Half (t1/2) for PF-07081532
Description: t1/2 is defined as the time measured for the plasma concentration to decrease by one half.
Time Frame: 0, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24 hours post-dose on Day 28 for Part A, on Day 42 for Part B and Part C
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part B | PF-07081532 180 mg Part C
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 12 | 9
hour | 26.50 (4.598) | 26.36 (6.265) | 23.68 (3.782) | 24.50 (5.442) | 20.70 (4.420) | 23.07 (5.855)

9. Secondary Outcome: Cumulative Amount of Drug Recovered Unchanged in Urine Over 24 Hours (Ae24) for PF-07081532
Description: Ae24 is defined as cumulative amount of drug recovered unchanged in urine over 24 hours using the method of urine concentration * volume of urine.
Time Frame: Part A: Day 28 (0-24 hours). Part C : Day 42 (0-24 hours)
Population: The population for this outcome measure included all randomized participants with T2DM who received at least 1 dose of PF-07081532 and had at least 1 of the PK parameters of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part C
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 6
mg |  |  |  | 0.1940 | 0.1054 (221)

10. Secondary Outcome: Percentage of Ae24 (Ae24%) for PF-07081532
Description: Ae24% is defined as percent of dose recovered unchanged in urine over the 24 hours using the method of 100 * Ae24/Dose
Time Frame: Part A: Day 28 (0-24 hours). Part C : Day 42 (0-24 hours)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Ae24
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part C
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 6
Percentage of Ae24 |  |  |  | 0.1620 | 0.05848 (221)

11. Secondary Outcome: Renal Clearance (CLr) for PF-07081532
Description: Renal clearance was calculated as cumulative amount of drug recovered unchanged in urine over the dosing interval tau (Aetau) divided by area under the concentration time-curve from time 0 to time tau (AUCtau)
Time Frame: Part A: Day 28 (0-24 hours). Part C : Day 42 (0-24 hours)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour (L/hr)
Arm/Group | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | PF-07081532 180 mg Part C
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 6
liter per hour (L/hr) |  |  |  | 0.0002690 | 0.0001935 (129)

ADVERSE EVENTS:
Time Frame: From the first dose up to 28-35 days after last administration of study intervention (that is a maximum of 63 days from first dose for Part A and a maximum of 77 days from first dose for Part B and Part C)
Description: MedDRA 24.0 coding dictionary was applied for all AE tables. The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo Part A | PF-07081532 10 mg Part A | PF-07081532 30 mg Part A | PF-07081532 60 mg Part A | PF-07081532 120 mg Part A | Placebo Part B | PF-07081532 180 mg Part B | Placebo Part C | PF-07081532 180 mg Part C
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7 | 0/8 | 0/8 | 0/8 | 0/3 | 0/12 | 0/2 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 1/8 | 0/8 | 0/8 | 0/3 | 0/12 | 0/2 | 0/9
Other Adverse Events (participants affected / at risk) | 7/9 | 3/7 | 7/8 | 8/8 | 8/8 | 3/3 | 11/12 | 2/2 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Part A (N=9) | PF-07081532 10 mg Part A (N=7) | PF-07081532 30 mg Part A (N=8) | PF-07081532 60 mg Part A (N=8) | PF-07081532 120 mg Part A (N=8) | Placebo Part B (N=3) | PF-07081532 180 mg Part B (N=12) | Placebo Part C (N=2) | PF-07081532 180 mg Part C (N=9)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo Part A (N=9) | PF-07081532 10 mg Part A (N=7) | PF-07081532 30 mg Part A (N=8) | PF-07081532 60 mg Part A (N=8) | PF-07081532 120 mg Part A (N=8) | Placebo Part B (N=3) | PF-07081532 180 mg Part B (N=12) | Placebo Part C (N=2) | PF-07081532 180 mg Part C (N=9)
Bandaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1/7 | 0/7 | 0/7 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 5 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 4 | 2 | 6 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 4 | 2 | 4 | 1 | 5 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 3
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 4 | 5 | 1 | 7 | 1 | 8
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 3 | 1 | 3 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 4 | 2 | 3 | 0 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 2 | 1 | 4 | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 6 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 2 | 0 | 2 | 4 | 3 | 1 | 2 | 0 | 3
Mental impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT04305587/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04305587/SAP_001.pdf